CLINICAL TRIAL: NCT05136404
Title: An Open-Label, Randomized Study to Evaluate the Relative Bioavailability of Selpercatinib in 3 Formulations for Pediatric Use
Brief Title: A Relative Bioavailability Study of Selpercatinib (LY3527723) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Loxo Oncology, Inc. (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 17821; J2G-MC-JZJU (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-11-25; First posted 2021-11-29 (Actual); Results first posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-02

CONDITIONS: Healthy
MeSH Terms: interventions — selpercatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Selpercatinib Sequence A: (Experimental): Period 1: 20 milligram (mg) Selpercatinib capsule single oral dose administered orally on Day 1.
  Period 2: 20 mg per milliliter (mL) Selpercatinib Powder for Oral suspension (PFOS) single oral suspension dose on Day 8.
  Period 3: 20 mg/mL Selpercatinib Ready to Use (RTU) single oral suspension on Day 15.
  Interventions: Drug: Selpercatinib
- Selpercatinib Sequence B (Experimental): Period 1: 20 mg/mL Selpercatinib RTU single oral suspension on Day 1.
  Period 2: 20 mg Selpercatinib capsule single oral dose administered orally on Day 8.
  Period 3: 20 mg/mL PFOS single oral suspension dose on Day 15.
  Interventions: Drug: Selpercatinib
- Selpercatinib Sequence C (Experimental): Period 1: 20 mg/mL PFOS single oral suspension dose on Day 1.
  Period 2: 20 mg/mL Selpercatinib RTU single oral suspension on Day 8.
  Period 3: 20 mg Selpercatinib capsule single oral dose administered orally on Day 15.
  Interventions: Drug: Selpercatinib

INTERVENTIONS:
Drug: Selpercatinib — Administered orally
  Other Names: LY3527723; LOXO-292

SUMMARY:
The main purpose of this study is to compare the amount of selpercatinib that gets into the blood stream and how long it takes the body to get rid of it, when given as three different formulations in adult healthy participants. The information about any adverse effects experienced will be collected and the tolerability of selpercatinib will also be evaluated. The study may last up to 59 days including the 28 days of screening period.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, and vital signs
* Body mass index (BMI) within the range 18.0 to 35.0 kilograms per meter squared (kg/m²)

Exclusion Criteria:

* Have a history of allergic reactions to medications or food products
* Have a clinically significant abnormality of blood pressure and/or pulse rate as determined by the investigator
* Clinically significant abnormalities on ECG as determined by the investigator or prolongation of the QTcB or QTcF >450 msec at screening
* Have clinically significant active cardiovascular disease or history of myocardial infarction within 6 months prior to the planned start of selpercatinib
* Have a history or presence of cardiovascular, respiratory, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the investigational product; or of interfering with the interpretation of data. Appendectomy, splenectomy, and cholecystectomy are considered as acceptable
* Use of H2 blockers, proton pump inhibitors, and other drugs that affect selpercatinib exposure within 7 days of screening
* Are intending to use over-the-counter or prescription medication, including dietary supplements, within 14 days prior to dosing and until study discharge (apart from occasional acetaminophen (≤2 g/24 hours), hormonal contraception, or hormone replacement therapy)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2022-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- LabCorp CRU, Inc., Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Selpercatinib Sequence A:: Period 1: 20 milligram (mg) Selpercatinib capsule single oral dose administered orally on Day 1.
  Period 2: 20 mg per milliliter (mL) Selpercatinib Powder for Oral suspension (PFOS) single oral suspension dose on Day 8.
  Period 3: 20 mg/mL Selpercatinib Ready to Use (RTU) single oral suspension on Day 15.
  Selpercatinib: Administered orally
- Selpercatinib Sequence B: Period 1: 20 mg/mL Selpercatinib RTU single oral suspension on Day 1.
  Period 2: 20 mg Selpercatinib capsule single oral dose administered orally on Day 8.
  Period 3: 20 mg/mL PFOS single oral suspension dose on Day 15.
  Selpercatinib: Administered orally
- Selpercatinib Sequence C: Period 1: 20 mg/mL PFOS single oral suspension dose on Day 1.
  Period 2: 20 mg/mL Selpercatinib RTU single oral suspension on Day 8.
  Period 3: 20 mg Selpercatinib capsule single oral dose administered orally on Day 15.
  Selpercatinib: Administered orally
Period: Period 1
Arm/Group | Selpercatinib Sequence A: | Selpercatinib Sequence B | Selpercatinib Sequence C
Started | 14 | 14 | 14
Received atLeast One Dose of Study Drug | 14 | 14 | 14
Completed | 14 | 13 | 13
Not Completed | 0 | 1 | 1
Not completed — Adverse Event | 0 | 1 | 1
Period: Period 2
Arm/Group | Selpercatinib Sequence A: | Selpercatinib Sequence B | Selpercatinib Sequence C
Started | 14 | 13 | 13
Completed | 14 | 13 | 12
Not Completed | 0 | 0 | 1
Not completed — Inappropriate Behavior | 0 | 0 | 1
Period: Period 3
Arm/Group | Selpercatinib Sequence A: | Selpercatinib Sequence B | Selpercatinib Sequence C
Started | 14 | 13 | 12
Completed | 14 | 13 | 11
Not Completed | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of Selpercatinib.
Groups:
- 20 mg Selpercatinib: Participants were randomized to 1 of 3 treatment sequences and will receive single doses of 20 mg Selpercatinib on each of Days 1, 8, and 15 as either the RTU suspension, the PFOS, or the capsule.
  Sequence A: Period 1: 20 milligram (mg) Selpercatinib capsule single oral dose administered orally on Day 1. Period 2: 20 mg per milliliter (mL) Selpercatinib Powder for Oral suspension (PFOS) single oral suspension dose on Day 8. Period 3: 20 mg/mL Selpercatinib Ready to Use (RTU) single oral suspension on Day 15.
  Sequence B: Period 1: 20 mg/mL Selpercatinib RTU single oral suspension on Day 1. Period 2: 20 mg Selpercatinib capsule single oral dose administered orally on Day 8. Period 3: 20 mg/mL PFOS single oral suspension dose on Day 15.
  Sequence C: Period 1: 20 mg/mL PFOS single oral suspension dose on Day 1. Period 2: 20 mg/mL Selpercatinib RTU single oral suspension on Day 8. Period 3: 20 mg Selpercatinib capsule single oral dose administered orally on Day 15.
Arm/Group | 20 mg Selpercatinib
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.0 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Selpercatinib
Description: PK: Cmax of Selpercatinib
Time Frame: Days 1, 8, and 15: Predose, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, and 144 hours (h) postdose
Population: All participants who received at least one dose of Selpercatinib and have evaluable pharmacokinetic (PK) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- 20 mg Selpercatinib Capsule (Reference): 20 mg Selpercatinib capsule administered orally.
- 20 mg Selpercatinib RTU Suspension (Test): 20 mg/mL Selpercatinib RTU administered orally.
- 20 mg/mL PFOS (Test): 20 mg/mL PFOS administered orally.
Arm/Group | 20 mg Selpercatinib Capsule (Reference) | 20 mg Selpercatinib RTU Suspension (Test) | 20 mg/mL PFOS (Test)
Number analyzed (Participants) | 38 | 41 | 41
nanograms per milliliter (ng/mL) | 176 (64.2) | 174 (36.9) | 180 (39.8)
Statistical Analysis 1: Comparison: 20 mg Selpercatinib Capsule (Reference) vs 20 mg Selpercatinib RTU Suspension (Test); Test type: Other; Mixed Models Analysis; Ratio of Geometric Least Squares Mean = 1.00, 90% CI 2-sided [0.937 to 1.08]
Statistical Analysis 2: Comparison: 20 mg Selpercatinib Capsule (Reference) vs 20 mg/mL PFOS (Test); Test type: Other; Mixed Models Analysis; Ratio of Geometric Least Squares Mean = 1.04, 90% CI 2-sided [0.968 to 1.11]

2. Primary Outcome: PK: Area Under the Plasma Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of Selpercatinib
Description: PK AUC[0-∞] of Selpercatinib
Time Frame: Days 1, 8, and 15: Predose, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, and 144 h postdose
Population: All participants who received at least one dose of selpercatinib and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | 20 mg Selpercatinib Capsule (Reference) | 20 mg Selpercatinib RTU Suspension (Test) | 20 mg/mL PFOS (Test)
Number analyzed (Participants) | 36 | 41 | 40
nanogram*hour per milliliter (ng*hr/mL) | 2540 (28.0) | 2410 (29.0) | 2490 (27.0)
Statistical Analysis 1: Comparison: 20 mg Selpercatinib Capsule (Reference) vs 20 mg Selpercatinib RTU Suspension (Test); Test type: Other; Mixed Models Analysis; Ratio of Geometric Least Squares Mean = 0.989, 90% CI 2-sided [0.953 to 1.03]
Statistical Analysis 2: Comparison: 20 mg Selpercatinib Capsule (Reference) vs 20 mg/mL PFOS (Test); Test type: Other; Mixed Models Analysis; Ratio of Geometric Least Squares Mean = 1.02, 90% CI 2-sided [0.982 to 1.06]

3. Primary Outcome: PK: Area Under the Plasma Concentration Versus Time Curve From Time Zero to the Last Measured Concentration Value (AUC[0-tlast]) of Selpercatinib
Description: PK: AUC[0-tlast] of Selpercatinib
Time Frame: Days 1, 8, and 15: Predose, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, and 144 h postdose
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | 20 mg Selpercatinib Capsule (Reference) | 20 mg Selpercatinib RTU Suspension (Test) | 20 mg/mL PFOS (Test)
Number analyzed (Participants) | 38 | 41 | 41
ng*hr/mL | 2180 (36.9) | 2160 (31.6) | 2190 (30.8)
Statistical Analysis 1: Comparison: 20 mg Selpercatinib Capsule (Reference) vs 20 mg Selpercatinib RTU Suspension (Test); Test type: Other; Mixed Models Analysis; Ratio of Geometric Least Squares Mean = 1.01, 90% CI 2-sided [0.972 to 1.06]
Statistical Analysis 2: Comparison: 20 mg Selpercatinib Capsule (Reference) vs 20 mg/mL PFOS (Test); Test type: Other; Mixed Models Analysis; Ratio of Geometric Least Squares Mean = 1.03, 90% CI 2-sided [0.992 to 1.08]

4. Primary Outcome: PK: Time to Maximum Observed Concentration (Tmax) of Selpercatinib
Description: PK: Tmax of Selpercatinib
Time Frame: Days 1, 8, and 15: Predose, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, and 144 h postdose
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Median (Full Range); unit: h
Arm/Group | 20 mg Selpercatinib Capsule (Reference) | 20 mg Selpercatinib RTU Suspension (Test) | 20 mg/mL PFOS (Test)
Number analyzed (Participants) | 38 | 41 | 41
h | 1.50 [1.00 to 24.02] | 1.50 [1.00 to 3.00] | 1.50 [1.00 to 3.50]
Statistical Analysis 1: Comparison: 20 mg Selpercatinib Capsule (Reference) vs 20 mg Selpercatinib RTU Suspension (Test); Test type: Superiority; p = 0.4728, Sign test; Median Difference (Final Values) = 0.00, 90% CI 2-sided [-0.50 to 0.00]
Statistical Analysis 2: Comparison: 20 mg Selpercatinib Capsule (Reference) vs 20 mg/mL PFOS (Test); Test type: Superiority; p = 0.0142, Sign test; Median Difference (Final Values) = 0.00, 90% CI 2-sided [-0.50 to 0.00]

ADVERSE EVENTS:
Time Frame: Baseline up to 59 days
Description: All enrolled participants who received at least one dose of selpercatinib, whether or not they completed all protocol requirements.
Groups:
- Selpercatinib Sequence B:: Period 1: 20 mg/mL Selpercatinib RTU single oral suspension on Day 1.
  Period 2: 20 mg Selpercatinib capsule single oral dose administered orally on Day 8.
  Period 3: 20 mg/mL PFOS single oral suspension dose on Day 15.
- Selpercatinib Sequence C:: Period 1: 20 mg/mL PFOS single oral suspension dose on Day 1.
  Period 2: 20 mg/mL Selpercatinib RTU single oral suspension on Day 8.
  Period 3: 20 mg Selpercatinib capsule single oral dose administered orally on Day 15.
Arm/Group | Selpercatinib Sequence A: | Selpercatinib Sequence B: | Selpercatinib Sequence C:
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/41 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/41 | 0/41
Other Adverse Events (participants affected / at risk) | 0/39 | 0/41 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-11-22): https://cdn.clinicaltrials.gov/large-docs/04/NCT05136404/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-09): https://cdn.clinicaltrials.gov/large-docs/04/NCT05136404/SAP_001.pdf